CLINICAL TRIAL: NCT06126575
Title: A Phase 1, Open-Label, Non-randomized, Parallel-Group Study to Evaluate the Pharmacokinetics, Safety and Tolerability of a Single Oral Dose of 200 mg Elacestrant in Subjects With Normal Hepatic Function or Severe Hepatic Impairment
Brief Title: A PK Study Testing Single Oral Dose of Elacestrant in Subjects With Normal or Severely Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STML-ELA-1023
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Hepatic Impairment
Keywords: metastatic breast cancer; breast cancer; elacestrant
MeSH Terms: conditions — Breast Neoplasms | interventions — RAD1901

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Subjects with normal hepatic function (Experimental): Subjects with normal hepatic function will receive treatment compared to subjects with severe hepatic function
  Interventions: Drug: Elacestrant dihydrochloride
- Subjects with severe hepatic impaired function (Experimental): Subjects with severe hepatic function will receive treatment compared to subjects with normal hepatic function
  Interventions: Drug: Elacestrant dihydrochloride

INTERVENTIONS:
Drug: Elacestrant dihydrochloride — A single oral dose of 200 mg elacestrant (2 x 100 mg tablets).

SUMMARY:
This is a Phase 1, multi-center, open-label, non-randomized, parallel group study to evaluate the effect of severe hepatic impairment on the PK, safety and tolerability of a single oral dose of Elacestrant.

DETAILED DESCRIPTION:
A total of 16 subjects will be recruited and divided between the following two Groups:

Group 1: 8 subjects with severe hepatic impairment Group 2: 8 subjects with normal hepatic function (control group)

On Day 1, subjects will receive a single oral dose of 200 mg Elacestrant (2 x 100 mg tablets). Safety assessment and blood sampling for Elacestrant analysis on plasma will be performed at predefined time points up to 240 hours post.

The total duration of study participation for each subject (from screening to the follow up call) is anticipated to be approximately 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the study procedures in the informed consent form (ICF) and be willing and able to comply with the protocol restrictions and requirements.
2. Males and Females older than 18 years.
3. Body mass index between 18.0 and 40.0 kg/m^2, inclusive.
4. Females must have non-functioning ovaries defined as postmenopausal and/or bilateral salpingo - oophorectomy. All female subjects must have a negative pregnancy test at screening and at check-in.
5. Males who are non-sterilized and sexually active with a female partner of childbearing potential must agree to use highly effective contraception from admission and for 120 days after IMP dose.
6. Males must agree not to donate sperm from admission and for 120 days after investigational medicinal product dose.
7. Non-smoker or light smoker, i.e. no more than 10 cigarettes or 10 mg equivalent use of Nicotine per day by e-vapor cigarette, pipe, cigar, chewing tobacco, nicotine patch, nicotine gum, AND able or willing to refrain from smoking and tobacco use for 2 hours prior to dose and 4 hours after IMP dose.

   Additional inclusion criteria applicable to subjects with Normal Hepatic Function Only
8. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations. NOTE: Congenital nonhemolytic hyperbilirubinemia/Gilbert's syndrome based on total and direct bilirubin is not acceptable.
9. Matched to subjects with severe hepatic impairment in gender, age (±10 years), weight (±10 kg) and race.

   Additional inclusion criteria applicable to subjects with Severe Hepatic Impairment Only
10. Documented chronic stable severe liver disease according to Child Pugh (CP) classification (CP score C) with diagnosis of hepatic impairment due to parenchymal liver disease. This will exclude biliary liver cirrhosis or other causes of hepatic impairment not related to parenchymal disorder.

    * 'Documented' is defined by medical history and physical examination, and confirmed by at least 1 of the following: hepatic ultrasound, computed axial tomography scan, magnetic resonance imaging, and/or liver biopsy.
    * 'Chronic' is defined as >6 months.
    * 'Stable' is defined as no clinically significant change in disease status within the last 6 weeks, as documented by the subject's recent medical history (eg, no worsening of clinical signs of hepatic impairment, or no worsening of total bilirubin or prothrombin time by more than 50%).
11. Subjects with severe hepatic impairment may have medical findings consistent with their hepatic dysfunction as determined by medical history, physical examination, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations at screening and check-in (Day -1), as assessed by the Investigator, provided that the followings are satisfied:

    * Non-hepatic impairment-related, abnormal clinical laboratory evaluations must not be clinically relevant, as judged by the Investigator and approved by the study assigned medical monitor.
    * Values outside the normal ranges for liver function tests are acceptable as consistent with the subject's hepatic condition, provided they are stable for at least 1 month prior to screening, as judged by the Investigator and approved by the study assigned medical monitor.
    * Subjects may enter with non-clinically significant Grade 1 anemia per CTCAE version 5.0, i.e. with Hb > 10 mg/dL.
    * Subjects must have a platelet count ≥ 35 × 109 /L
12. Subjects with stable, mild, chronic concurrent diseases, such as degenerative joint disease, hypertension or hyperlipidaemia, etc. may be included. Subjects with diabetes mellitus may be included, provided the subjects have:

    * Glycosylated hemoglobin A1c values ≤ 9.5% at screening; eligibility in case of outside values should be evaluated by the study assigned medical monitor on a case-by-case basis.
    * Blood glucose values ≤ 240 mg/dL at screening and check-in (Day -1) while on subjects' normal diabetes medication.
13. Currently on a stable medication regimen, defined as not starting new drug(s) or changing drug dose(s) within 28 days of administration of study drug (Day 1). Concomitant medications administered within 28 days prior to administration of study drug (Day 1) must be approved by the Investigator and the study assigned medical monitor.

Exclusion Criteria:

1. Presence of any condition or circumstance that prevents the subject from understanding and signing the ICF.
2. Presence or history of any disorder that may prevent the successful completion of the study.
3. History of significant hypersensitivity, intolerance, or allergy to food, or any medical product or relevant excipient, unless approved by the Investigator.
4. History of allergy to Elacestrant or drugs in a similar pharmacology class (selective ER modulator or SERD) or excipients used in the formulations of these drugs.
5. History of stomach or intestinal surgery or resection, or any significant gastrointestinal disease (eg, Crohn's disease) that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed). Cholecystectomy will be allowed at the discretion of the Investigator.
6. Acute disease state (eg, nausea, vomiting, fever, diarrhea) within 14 days prior to check-in.
7. History of drug/chemical abuse within 1 year prior to check-in.
8. History of alcohol abuse within 3 months prior to screening and/or consume > 21 units per week for males and > 14 units for females. One unit of alcohol equals 12 oz (360 mL) beer, 1 1⁄2 oz (45 mL) liquor, or 5 oz (150 mL) wine.
9. Positive drug screen at screening, or positive alcohol or drug screen at check-in.
10. Participation in a clinical study involving administration of an investigational drug (new chemical entity) or device in the past 28 days or 5 half-lives (whichever is longer) prior to dosing.
11. Received Elacestrant within 60 days prior to dosing.
12. Corrected value of the interval between the Q and T waves on the ECG tracing, using Fridericia's formula, is > 450 ms (for healthy males) or > 470 ms (for healthy females), is > 470 ms (for hepatic impairment males) or > 480 ms (for hepatic impairment females); or has ECG findings deemed abnormal with clinical significance by the Investigator at screening. ECGs will be collected in triplicate.
13. Use of any drugs or herbal remedies known to be strong or moderate inhibitors or inducers of CYP3A enzymes for 28 days prior to dosing or 5 half-lives (whichever is longer) and throughout the study.
14. Not willing to follow on-study diet requirements.
15. Ingestion of Seville orange- or grapefruit- containing foods or beverages within 28 days prior to check-in.
16. Receipt of blood products within 2 months prior to check-in.
17. Donation of blood from 3 months prior to screening, plasma from 2 weeks prior to screening, or platelets from 6 weeks prior to screening.
18. Poor peripheral venous access.
19. Subjects who, in the opinion of the Investigator, should not participate in this study.

    Additional exclusion criteria applicable to Subjects with Normal Hepatic Function Only
20. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular (including any prior history of cardiomyopathy or cardiac failure), gastrointestinal, neurological, or psychiatric disorder.
21. Unable to refrain from or anticipate the use of any non-prescription medications, herbal remedies, or vitamin supplements within 14 days prior to dosing and throughout the study.

    NOTE: After check-in, acetaminophen (up to 2 g per 24 hours), and 1% hydrocortisone cream may be administered at the discretion of the Investigator.
22. Unable to refrain from or anticipate the use of any prescription medications within 28 days prior to dosing or 5 half-lives (whichever is longer) and throughout the study, unless approved by the Investigator and the study assigned medical monitor.

    NOTE: slow-release medications / products considered to still be active prior to check-in must be approved by the Investigator and the study assigned medical monitor.
23. Positive hepatitis B panel test and/or positive hepatitis C RNA test. Subjects whose results are compatible with prior immunization may be included.
24. History of diabetes mellitus.

    Additional exclusion criteria applicable to Subjects with Hepatic Impairment Only
25. Grade 3 and Grade 4 encephalopathy as determined by the CP score.
26. Portal systemic shunt.
27. Subject has shown evidence of hepatorenal syndrome or abnormal serum creatinine levels (above upper limit for the local lab) and estimated glomerular filtration rate < 60 mL/min or abnormal sodium and potassium levels. The determination of the severity and clinical relevance of the latter 2 abnormalities will be at the discretion of the Investigator.
28. Treatment for gastrointestinal bleeding within the 3 months prior to check-in.
29. New medication or a change in dose for hepatic encephalopathy within the 3 months prior to check-in, unless approved by the Investigator and the study assigned medical monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Predose 240 hours after drug administration
Area under the plasma concentration-time curve from time zero to the last measurable concentration (AUC0-t) | Predose 240 hours after drug administration
AUC from time zero to infinity (AUC0-∞) | Predose 240 hours after drug administration

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Inland Empire Clinical Trials, LLC, Yucaipa, California
  - Floridian Clinical Research, Miami, Florida
  - American Research Corp, San Antonio, Texas